CLINICAL TRIAL: NCT01322165
Title: National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions
Acronym: GenTAC
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1438; 268201000048C-5-0-1 (NIH); N01HV68199-7-0-1 (NIH)
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Marfan Syndrome; Turner Syndrome; Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome; FBN1, TGFBR1, TGFBR2, ACTA2 or MYH11 Genetic Mutation; Bicuspid Aortic Valve Without Known Family History; Bicuspid Aortic Valve With Family History; Bicuspid Aortic Valve With Coarctation; Familial Thoracic Aortic Aneurysm and Dissections; Shprintzen-Goldberg Syndrome; Other Aneur/Diss of Thoracic Aorta Not Due to Trauma, <50yo; Other Congenital Heart Disease
Keywords: Marfan syndrome; Turner syndrome; Bicuspid aortic valve; Ehlers-Danlos Syndrome; Loeys-Dietz syndrome; Aneurysm; Genetic; aortic; thoracic; mutation; dissection
MeSH Terms: conditions — Marfan Syndrome; Turner Syndrome; Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome; Colorectal Cancer, Hereditary Nonpolyposis, Type 6; Aortic Aneurysm, Familial Thoracic 1; Shprintzen Golberg craniosynostosis; Bicuspid Aortic Valve Disease; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If a blood specimen is obtained, it is separated and stored as plasma, viable cells, and extracted DNA. If a saliva specimen is obtained, it is stored for DNA.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions (GenTAC) was initiated in 2006 by the National Heart, Lung, and Blood Institute (NHLBI) and the National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS). GenTAC established a registry of 3706 patients with genetic conditions that may be related to thoracic aortic aneurysms and collected medical data and biologic samples. The study ended in September 2016. Data and samples are available from NHLBI and requests should be made to BioLINCC. See the NHLBI website for more information: https://www.nhlbi.nih.gov/research/resources/gentac/.

ELIGIBILITY:
Eligible subjects must have one of the conditions listed below and be enrolled in-person at one of the participating clinical centers.Contact the study coordinator at the location nearest you for more information about participation.

* Marfan syndrome
* Turner syndrome
* Ehlers-Danlos syndrome
* Loeys-Dietz syndrome
* FBN1, TGFBR1, TGFBR2, ACTA2 or MYH11 genetic mutation
* Bicuspid aortic valve without known family history
* Bicuspid aortic valve with family history
* Bicuspid aortic valve with coarctation
* Familial Thoracic Aortic Aneurysm and DissectionsYes
* Shprintzen-Goldberg syndrome
* Other aneurysms and dissections of the thoracic aorta not due to trauma, <50yo
* Other congenital heart disease (e.g., Tetralogy of Fallot, coarctation)

Exclusion Criteria:

* Inability of the patient, parent or guardian to give consent.
* Unwillingness to provide a blood or buccal specimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort consists of patients with conditions related to genetically-induced thoracic aortic aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 3706 (Actual)
Dates: Start 2007-11; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Thoracic aortic aneurysms and dissections and their associated surgical interventions | bi-annual

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kroner, PhD, MPH, Study Director — RTI International; Richard Devereux, MD, Principal Investigator — The New York Presbyterian Hospital-Weill Cornell Medical Center; William Ravekes, M.D., Principal Investigator — Johns Hopkins University; Reed E. Pyeritz, M.D., Ph.D., Principal Investigator — University of Pennsylvania; Dianna M. Milewicz, M.D. Ph.D., Principal Investigator — University of Texas Medical School at Houston; Scott A. LeMaire, M.D., Principal Investigator — Baylor College of Medicine; Cheryl L. Maslen, Ph.D., Principal Investigator — Oregon Health and Science University; Ralph Shohet, MD, Principal Investigator — University of Hawaii; Jennifer Habashi, MD, Principal Investigator — Johns Hopkins University; Federico M. Asch, MD,FACC,FASE, Principal Investigator — MedStar Health; Kim Eagle, M.D., Study Chair — University of Michigan
Locations (7):
- United States (7):
  - Queens Medical Center, Honolulu, Hawaii
  - Johns Hopkins University, Baltimore, Maryland
  - The New York Presbyterian Hospital-Weill Cornell Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Medical School at Houston, Houston, Texas

REFERENCES:
- [Background] Eagle KA; GenTAC Consortium. Rationale and design of the National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions (GenTAC). Am Heart J. 2009 Feb;157(2):319-26. doi: 10.1016/j.ahj.2008.10.005. Epub 2008 Dec 17. PMID 19185640
- [Background] Matt P, Schoenhoff F, Habashi J, Holm T, Van Erp C, Loch D, Carlson OD, Griswold BF, Fu Q, De Backer J, Loeys B, Huso DL, McDonnell NB, Van Eyk JE, Dietz HC; GenTAC Consortium. Circulating transforming growth factor-beta in Marfan syndrome. Circulation. 2009 Aug 11;120(6):526-32. doi: 10.1161/CIRCULATIONAHA.108.841981. Epub 2009 Jul 27. PMID 19635970
- [Background] Kuang SQ, Guo DC, Prakash SK, McDonald ML, Johnson RJ, Wang M, Regalado ES, Russell L, Cao JM, Kwartler C, Fraivillig K, Coselli JS, Safi HJ, Estrera AL, Leal SM, LeMaire SA, Belmont JW, Milewicz DM; GenTAC Investigators. Recurrent chromosome 16p13.1 duplications are a risk factor for aortic dissections. PLoS Genet. 2011 Jun;7(6):e1002118. doi: 10.1371/journal.pgen.1002118. Epub 2011 Jun 16. PMID 21698135
- [Background] Mendoza DD, Kochar M, Devereux RB, Basson CT, Min JK, Holmes K, Dietz HC, Milewicz DM, LeMaire SA, Pyeritz RE, Bavaria JE, Maslen CL, Song H, Kroner BL, Eagle KA, Weinsaft JW; GenTAC (National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions) Study Investigators. Impact of image analysis methodology on diagnostic and surgical classification of patients with thoracic aortic aneurysms. Ann Thorac Surg. 2011 Sep;92(3):904-12. doi: 10.1016/j.athoracsur.2011.03.130. Epub 2011 Jul 2. PMID 21723533
- [Background] LeMaire SA, McDonald ML, Guo DC, Russell L, Miller CC 3rd, Johnson RJ, Bekheirnia MR, Franco LM, Nguyen M, Pyeritz RE, Bavaria JE, Devereux R, Maslen C, Holmes KW, Eagle K, Body SC, Seidman C, Seidman JG, Isselbacher EM, Bray M, Coselli JS, Estrera AL, Safi HJ, Belmont JW, Leal SM, Milewicz DM. Genome-wide association study identifies a susceptibility locus for thoracic aortic aneurysms and aortic dissections spanning FBN1 at 15q21.1. Nat Genet. 2011 Sep 11;43(10):996-1000. doi: 10.1038/ng.934. PMID 21909107
- [Background] Guo DC, Regalado E, Casteel DE, Santos-Cortez RL, Gong L, Kim JJ, Dyack S, Horne SG, Chang G, Jondeau G, Boileau C, Coselli JS, Li Z, Leal SM, Shendure J, Rieder MJ, Bamshad MJ, Nickerson DA; GenTAC Registry Consortium; National Heart, Lung, and Blood Institute Grand Opportunity Exome Sequencing Project; Kim C, Milewicz DM. Recurrent gain-of-function mutation in PRKG1 causes thoracic aortic aneurysms and acute aortic dissections. Am J Hum Genet. 2013 Aug 8;93(2):398-404. doi: 10.1016/j.ajhg.2013.06.019. Epub 2013 Aug 1. PMID 23910461
- [Background] Prakash S, Guo D, Maslen CL, Silberbach M, Milewicz D, Bondy CA; GenTAC Investigators. Single-nucleotide polymorphism array genotyping is equivalent to metaphase cytogenetics for diagnosis of Turner syndrome. Genet Med. 2014 Jan;16(1):53-9. doi: 10.1038/gim.2013.77. Epub 2013 Jun 6. PMID 23743550
- [Background] Cook JR, Carta L, Benard L, Chemaly ER, Chiu E, Rao SK, Hampton TG, Yurchenco P; GenTAC Registry Consortium; Costa KD, Hajjar RJ, Ramirez F. Abnormal muscle mechanosignaling triggers cardiomyopathy in mice with Marfan syndrome. J Clin Invest. 2014 Mar;124(3):1329-39. doi: 10.1172/JCI71059. Epub 2014 Feb 17. PMID 24531548
- [Background] Song HK, Preiss LR, Maslen CL, Kroner B, Devereux RB, Roman MJ, Holmes KW, Tolunay HE, Desvigne-Nickens P, Asch FM, Milewski RK, Bavaria J, LeMaire SA; GenTAC Consortium. Valve-sparing aortic root replacement in patients with Marfan syndrome enrolled in the National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions. J Heart Valve Dis. 2014 May;23(3):292-8. PMID 25296451
- [Background] Doyle JJ, Doyle AJ, Wilson NK, Habashi JP, Bedja D, Whitworth RE, Lindsay ME, Schoenhoff F, Myers L, Huso N, Bachir S, Squires O, Rusholme B, Ehsan H, Huso D, Thomas CJ, Caulfield MJ, Van Eyk JE, Judge DP, Dietz HC; GenTAC Registry Consortium; MIBAVA Leducq Consortium. A deleterious gene-by-environment interaction imposed by calcium channel blockers in Marfan syndrome. Elife. 2015 Oct 27;4:e08648. doi: 10.7554/eLife.08648. PMID 26506064
- [Background] Asch FM, Yuriditsky E, Prakash SK, Roman MJ, Weinsaft JW, Weissman G, Weigold WG, Morris SA, Ravekes WJ, Holmes KW, Silberbach M, Milewski RK, Kroner BL, Whitworth R, Eagle KA, Devereux RB, Weissman NJ; GenTAC Investigators. The Need for Standardized Methods for Measuring the Aorta: Multimodality Core Lab Experience From the GenTAC Registry. JACC Cardiovasc Imaging. 2016 Mar;9(3):219-26. doi: 10.1016/j.jcmg.2015.06.023. Epub 2016 Feb 17. PMID 26897684
- [Background] Guo DC, Gong L, Regalado ES, Santos-Cortez RL, Zhao R, Cai B, Veeraraghavan S, Prakash SK, Johnson RJ, Muilenburg A, Willing M, Jondeau G, Boileau C, Pannu H, Moran R, Debacker J; GenTAC Investigators, National Heart, Lung, and Blood Institute Go Exome Sequencing Project; Montalcino Aortic Consortium; Bamshad MJ, Shendure J, Nickerson DA, Leal SM, Raman CS, Swindell EC, Milewicz DM. MAT2A mutations predispose individuals to thoracic aortic aneurysms. Am J Hum Genet. 2015 Jan 8;96(1):170-7. doi: 10.1016/j.ajhg.2014.11.015. Epub 2014 Dec 31. PMID 25557781
- [Background] Kuang SQ, Medina-Martinez O, Guo DC, Gong L, Regalado ES, Reynolds CL, Boileau C, Jondeau G, Prakash SK, Kwartler CS, Zhu LY, Peters AM, Duan XY, Bamshad MJ, Shendure J, Nickerson DA, Santos-Cortez RL, Dong X, Leal SM, Majesky MW, Swindell EC, Jamrich M, Milewicz DM. FOXE3 mutations predispose to thoracic aortic aneurysms and dissections. J Clin Invest. 2016 Mar 1;126(3):948-61. doi: 10.1172/JCI83778. Epub 2016 Feb 8. PMID 26854927
- [Background] Prakash S, Kuang SQ; GenTAC Registry Investigators; Regalado E, Guo D, Milewicz D. Recurrent Rare Genomic Copy Number Variants and Bicuspid Aortic Valve Are Enriched in Early Onset Thoracic Aortic Aneurysms and Dissections. PLoS One. 2016 Apr 19;11(4):e0153543. doi: 10.1371/journal.pone.0153543. eCollection 2016. PMID 27092555
- [Background] Weinsaft JW, Devereux RB, Preiss LR, Feher A, Roman MJ, Basson CT, Geevarghese A, Ravekes W, Dietz HC, Holmes K, Habashi J, Pyeritz RE, Bavaria J, Milewski K, LeMaire SA, Morris S, Milewicz DM, Prakash S, Maslen C, Song HK, Silberbach GM, Shohet RV, McDonnell N, Hendershot T, Eagle KA, Asch FM; GENTAC Registry Investigators. Aortic Dissection in Patients With Genetically Mediated Aneurysms: Incidence and Predictors in the GenTAC Registry. J Am Coll Cardiol. 2016 Jun 14;67(23):2744-2754. doi: 10.1016/j.jacc.2016.03.570. PMID 27282895
- [Background] Roman MJ, Pugh NL, Hendershot TP, Devereux RB, Dietz H, Holmes K, Eagle KA, LeMaire SA, Milewicz DM, Morris SA, Pyeritz RE, Ravekes WJ, Shohet RV, Silberbach M; GenTAC InvestigatorsDietzHarry C.HabashiJenniferPrakashSiddharth K.MaslenCheryl L.SongHoward K.BavariaJoseph E.MilewskiKariannaWeinsaftJonathan W.McDonnellNazliAschFederico M.TolunayH. EserDesvigne-NickensPatriceTsengHungKronerBarbara L. Aortic Complications Associated With Pregnancy in Marfan Syndrome: The NHLBI National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions (GenTAC). J Am Heart Assoc. 2016 Aug 11;5(8):e004052. doi: 10.1161/JAHA.116.004052. PMID 27515814
- [Background] Prakash SK, Bondy CA, Maslen CL, Silberbach M, Lin AE, Perrone L, Limongelli G, Michelena HI, Bossone E, Citro R; BAVCon Investigators, GenTAC Registry Investigators; Lemaire SA, Body SC, Milewicz DM. Autosomal and X chromosome structural variants are associated with congenital heart defects in Turner syndrome: The NHLBI GenTAC registry. Am J Med Genet A. 2016 Dec;170(12):3157-3164. doi: 10.1002/ajmg.a.37953. Epub 2016 Sep 8. PMID 27604636
- [Background] Guo DC, Grove ML, Prakash SK, Eriksson P, Hostetler EM, LeMaire SA, Body SC, Shalhub S, Estrera AL, Safi HJ, Regalado ES, Zhou W, Mathis MR; GenTAC Investigators; BAVCon Investigators; Eagle KA, Yang B, Willer CJ, Boerwinkle E, Milewicz DM. Genetic Variants in LRP1 and ULK4 Are Associated with Acute Aortic Dissections. Am J Hum Genet. 2016 Sep 1;99(3):762-769. doi: 10.1016/j.ajhg.2016.06.034. Epub 2016 Aug 25. PMID 27569546
- [Result] Song HK, Bavaria JE, Kindem MW, Holmes KW, Milewicz DM, Maslen CL, Pyeritz RE, Basson CT, Eagle K, Tolunay HE, Kroner BL, Dietz H, Menashe V, Devereux RB, Desvigne-Nickens P, Ravekes W, Weinsaft JW, Brambilla D, Stylianou MP, Hendershot T, Mitchell MS, LeMaire SA; National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions (GenTAC) Consortium. Surgical treatment of patients enrolled in the national registry of genetically triggered thoracic aortic conditions. Ann Thorac Surg. 2009 Sep;88(3):781-7; discussion 787-8. doi: 10.1016/j.athoracsur.2009.04.034. PMID 19699898
- [Result] Kroner BL, Tolunay HE, Basson CT, Pyeritz RE, Holmes KW, Maslen CL, Milewicz DM, LeMaire SA, Hendershot T, Desvigne-Nickens P, Devereux RB, Dietz HC, Song HK, Ringer D, Mitchell M, Weinsaft JW, Ravekes W, Menashe V, Eagle KA. The National Registry of Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions (GenTAC): results from phase I and scientific opportunities in phase II. Am Heart J. 2011 Oct;162(4):627-632.e1. doi: 10.1016/j.ahj.2011.07.002. PMID 21982653
- [Result] Song HK, Kindem M, Bavaria JE, Dietz HC, Milewicz DM, Devereux RB, Eagle KA, Maslen CL, Kroner BL, Pyeritz RE, Holmes KW, Weinsaft JW, Menashe V, Ravekes W, LeMaire SA; Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions Consortium. Long-term implications of emergency versus elective proximal aortic surgery in patients with Marfan syndrome in the Genetically Triggered Thoracic Aortic Aneurysms and Cardiovascular Conditions Consortium Registry. J Thorac Cardiovasc Surg. 2012 Feb;143(2):282-6. doi: 10.1016/j.jtcvs.2011.10.024. Epub 2011 Nov 20. PMID 22104675
- [Result] Holmes KW, Maslen CL, Kindem M, Kroner BL, Song HK, Ravekes W, Dietz HC, Weinsaft JW, Roman MJ, Devereux RB, Pyeritz RE, Bavaria J, Milewski K, Milewicz D, LeMaire SA, Hendershot T, Eagle KA, Tolunay HE, Desvigne-Nickens P, Silberbach M; GenTAC Registry Consortium. GenTAC registry report: gender differences among individuals with genetically triggered thoracic aortic aneurysm and dissection. Am J Med Genet A. 2013 Apr;161A(4):779-86. doi: 10.1002/ajmg.a.35836. Epub 2013 Feb 26. PMID 23444191
- See also: GenTAC project resources being maintained by NHLBI since contract end. — https://www.nhlbi.nih.gov/research/resources/gentac/